CLINICAL TRIAL: NCT05850910
Title: Comparison Of The Immediate Effects Of Manipulation On The Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Approval Number: 19.01.2023-29
Record Dates: First submitted 2023-04-30; First posted 2023-05-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Vagus Nerve Autonomic Disorder
Keywords: manipulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine practice group (Experimental): The participant was asked to cross his arms in front of his body while lying on his back.
  Interventions: Other: Supine practice group
- Prone application group (Experimental): The participant positions their hands freely from the side of the treatment table in the prone position.
  Interventions: Other: Prone application group

INTERVENTIONS:
Other: Supine practice group — The practitioner's arm was placed in the mid-thoracic region from the opposite side of the individual's torso in the form of a half fist. In this position, the SPs coincide with the space in the middle of the half fist, while the TPs coincide with the fingertips and the thenar region. With the practitioner's other hand supporting the patient's elbows, a high-speed-low-amplitude thrust is applied from front to back.
  Arms: Supine practice group
Other: Prone application group — the practitioner positions the hypothenar part of his hands above the TPs in the mid-thoracic segment. From this point, a high-velocity-low-amplitude thrust is applied from the back to the front.
  Arms: Prone application group

SUMMARY:
High velocity low amplitude thrust applied at the vertebral level during spinal manipulation is thought to slide the vertebrae over each other and alter segmental biomechanics.

DETAILED DESCRIPTION:
Evidence suggests that spinal HVLA techniques may produce acute changes in skin sympathetic nerve activity. There are studies reporting that thoracic HVLA manipulation causes a statistically significant increase in cardiac vagal activity in the immediate post-intervention period compared to sham administration.

ELIGIBILITY:
Inclusion criteria:

* People who volunteered to work and signed the consent form
* Not having any of the application contraindications or exclusion criteria.
* Being between the ages of 18-45

Exclusion criteria:

* Presence of tumor, infection, trauma, inflammation
* Neurological problems (Acute myelopathy, spinal cord compression, cauda equina syndrome, nerve root compression)
* Vascular disorders (Vertebrobasilar insufficiency or cervical artery abnormalities, aortic aneurysm, angina pectoris, acute abdominal pain with preservation)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system device | one day
  The Polar H10 device is a heart rate sensor that comes with a wearable chest strap and is the gold standard of high sensitivity and accuracy. It can be connected to multiple training devices via Bluetooth and ANT+. The device comes with a soft, adjustable sensor that touches the chest to capture the heart rate in real time.
  In the study, the autonomic nervous system will be evaluated with the Polar H10 device. By connecting the device to a smart phone via bluetooth, the data will be recorded and the software supported by the device will be used for the analysis of the data.
Finger Oximeter | one day
  Finger oximeter (finger pulse oximeter) measures heart rate per minute and oxygen level in blood easily and quickly.
  This device, which is placed on the fingertip, measures the oxygen saturation by sensing the color tone changes in the blood depending on the oxygen with infrared rays. Oxygen saturation refers to the oxygen saturation in the blood. Typical oxygen saturation levels in a healthy person range from 95-100%. In people with lung problems, these values may be slightly lower.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Rodrigues PTV, Correa LA, Reis FJJ, Meziat-Filho NA, Silva BM, Nogueira LAC. One Session of Spinal Manipulation Improves the Cardiac Autonomic Control in Patients with Musculoskeletal Pain: A Randomized Placebo-Controlled Trial. Spine (Phila Pa 1976). 2021 Jul 15;46(14):915-922. doi: 10.1097/BRS.0000000000003962. PMID 33496535